CLINICAL TRIAL: NCT05114915
Title: Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of Docetaxel for Injection (Albumin-bound) in Different Dose Regimens in Patients With Advanced Solid Tumors: An Open-label, Multicenter, Phase 1b Study
Brief Title: A Study to Evaluate the Safety and Efficacy of Docetaxel for Injection (Albumin-bound)in Different Dose Regimens in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB1801-CSP-004
Record Dates: First submitted 2021-10-12; First posted 2021-11-10 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-10

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Docetaxel for Injection-qw 3/4 regimen (Experimental): Docetaxel for Injection (Albumin-bound) will be administrated once every week in the first three weeks (Day 1, 8 and 15) in every 28-day cycle, starting at a dose of 30 mg/m^2.
  Interventions: Drug: Albumin-bound docetaxel
- Docetaxel for Injection-q2w 2/4 regimen (Experimental): Docetaxel for Injection (Albumin-bound) will be administrated once every week every other week (Day 1 and 15) in every 28-day cycle, starting at a dose of 50 mg/m^2.
  Interventions: Drug: Albumin-bound docetaxel
- Docetaxel for Injection-qw 2/3 regimen (Experimental): Docetaxel for Injection (Albumin-bound) will be administrated once every week in the first two weeks (Day 1 and 8) in every 21-day cycle, starting at a dose of 30 mg/m^2.
  Interventions: Drug: Albumin-bound docetaxel

INTERVENTIONS:
Drug: Albumin-bound docetaxel — Albumin-bound docetaxel by intravenous infusion

SUMMARY:
The aim of this study is designed to evaluate the safety, tolerability, pharmacokinetics and preliminary antitumor activity of docetaxel for injection (albumin-bound) in different dose regimens in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study will be conducted in two stages. The first stage (Stage I) is a dose-escalation study. A classic 3+3 design will be used to determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D). Patients will receive the docetaxel for injection (albumin-bound) until disease progression, or intolerable toxicity, or other reasons for termination of the study. All dose-escalation decisions will be based on the safety data generated from the current highest dose group.

In the cohort-expansion study (Stage Ⅱ), patients with a potential to have better response to the study drug will be recruited. Patients will receive the docetaxel for injection (albumin-bound) at the recommended phase 2 dose (RP2D) and follow the treatment regimen established in Stage I.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18, ≤75 years (subject to the date when the informed consent form is signed) and voluntarily signed the informed consent form.
2. Histologically or cytologically confirmed diagnosis of advanced or metastatic solid tumors, for which standard therapy either does not exist or has proven to be ineffective, intolerable or unacceptable for the patient.
3. At least one measurable lesion according to RECISTv1.1.
4. Patients with Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
5. Patients with estimated survival time of ≥ 3 months.
6. Main organ function meets the following criteria within 7 days before treatment (no medical supportive treatments such as blood component transfusion, human granulocyte colony-stimulating factor (G-CSF), thrombopoietin (TPO), interleukin-11, and erythropoietin (EPO) within 2 weeks before baseline examination):

   Absolute neutrophil count ≥1.5×10^9/L; Platelets ≥100×10^9/L; Hemoglobin ≥90 g/L or ≥5.6 mmol/L; Serum creatinine ≤ 1.5×ULN or creatinine clearance rate ≥ 50 mL/min; Liver function: total bilirubin≤ 1.0 × ULN, ≤ 1.5 × ULN for patients with liver metastasis or liver cancer; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN, ≤ 2.5 × ULN for patients with liver metastasis or liver cancer.
7. Fertile patients must use contraceptive measures (such as intrauterine device [IUD], contraceptive pill or condom) during the study period and within 6 months after the end of the study, and men should avoid sperm donation; Women of childbearing age must have negative serum pregnancy test within 7 days before study enrollment, and must be non-lactating women.

Exclusion Criteria:

1. Patients with central nervous system metastasis or meningeal metastasis, accompanied by the following conditions:

1. Patients with clinical symptoms related to central nervous system metastasis or meningeal metastasis;
2. New lesions in the brain or progression of the original lesions on imaging from the end of brain radiotherapy or surgery to the first administration;
3. Central nervous system metastasis with cortical alcohols, radiotherapy, dehydration drugs and other drugs for symptoms control within the last two weeks;
4. Patients has brain stem (midbrain, pons, medulla oblongata) metastasis;
5. Other evidence shows that the patient's central nervous system metastasis or meningeal metastasis has not been controlled, which is not suitable for inclusion according to the judgment of the researcher.

2. Known human immunodeficiency virus (HIV) test positive or known history of acquired immunodeficiency syndrome (AIDS), history of organ transplantation, history of serious autoimmune diseases judged by the researchers to be unsuitable for inclusion.

3. HCV antibody (+) or active hepatitis B (HBsAg positive and HBV DNA > 500 IU/mL) and uncontrolled active infection (those who must receive systematic anti infection treatment, or those with unexplained body temperature > 38 ℃ (axillary temperature) before administration).

4. Patients have a history of serious cardiovascular diseases, including but not limited to:

1. Severe heart rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention and third-degree atrioventricular block;
2. History of myocardial infarction, angina pectoris, angioplasty, coronary artery bypass surgery;
3. Patients with prolonged QT/QTc interval (QTcF > 480 ms, Fridericia's formula: QTcF = QT/RR^0.33, RR = 60/heart rate) by ECG during the screening period;
4. left ventricular ejection fraction (LVEF) ≤ 50% by echocardiography (ECHO) or multi-gated acquisition (MUGA) during the screening period;
5. Heart failure with New York Heart Association (NYHA) Classification of Class Ш and above;
6. Poorly controlled hypertension (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 95 mmHg despite optimal treatment);
7. Previous or current cardiomyopathy;
8. Patients with severe pulmonary hypertension or a history of pulmonary embolism within 6 months.

5. Patients with a third space effusion (e.g., pleural effusion, ascites, or pericardial effusion) that is difficult to control, who, in the judgment of the investigator, are not suitable for the study.

6. Allergic history to taxane or any excipients of the study drug (CTCAE 5.0 grade ≥ 3 grade).

7. Adverse reactions from the previous anti-tumor treatment have not yet recovered to ≤ level 1 based on CTCAE 5.0 (except for the toxicity without safety risk judged by the investigator, such as alopecia).

8. Patients who have previously received docetaxel containing regimen and progressed during treatment or within 6 months after treatment.

9. Patients who have undergone major organ surgery (excluding puncture biopsy) or significant trauma within 4 weeks before the first dose of the investigational drug, or who need to undergo elective surgery during the study period.

10. The time between the last anti-tumor treatment and the first medication meet the following time interval: anti-tumor treatment such as chemotherapy, radiotherapy (except local radiotherapy for pain relief), targeted therapy, immunotherapy and other clinical research drugs within 4 weeks before the first administration; oral fluorouracils, small molecule targeted drugs and traditional Chinese medicine with anti-tumor indications within 2 weeks before the first administration.

11. Patients who have received corticosteroid (prednisone > 10 mg/day or equivalent) or other immunosuppressive therapies within 2 weeks before the first dose of the investigational drug, except for the following: a. use of topical, ocular, intra-articular, nasal and inhaled glucocorticoids; b. short-term use of glucocorticoids for prophylaxis (such as prevention of contrast agent allergy).

12. Patients who have used potent inhibitors or inducers of CYP3A4 within 2 weeks before the first dose of the investigational drug.

13. Patients with alcohol or drug dependence. 14. Patients have clear history of neurological or psychiatric disorders, including epilepsy and dementia.

15. The researcher believes that the patient has other reasons that affect the safety or compliance, or is not in the best interests of the subject and is not suitable to participate in this clinical study (for example, eye diseases, venous thrombosis, etc., which affect the safety according to the judgment of the researcher).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The occurrence and frequency of adverse events and serious adverse events | Up to approximately 2 years
  Incidence of adverse events and serious adverse events
The maximum tolerated dose (MTD) (if available) and recommended phase 2 dose (RP2D) in stage I | At the end of Cycle 1 (each cycle is 28 or 21 days)
  The maximum tolerated dose
Overall response rate (ORR) in stage Ⅱ | Up to approximately 2 years
  Objective response rate
Progression-free survival (PFS) in stage Ⅱ | Up to approximately 2 years
  Progression-free survival
Disease control rate (DCR) in stage Ⅱ | Up to approximately 2 years
  Disease control rate
Duration of response (DOR) in stage Ⅱ | Up to approximately 2 years
  Duration of response

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration (AUC0-last) | At the end of Cycle 1 (each cycle is 28 or 21 days)
  Area under the plasma concentration-time curve
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) | At the end of Cycle 1 (each cycle is 28 or 21 days)
  Area under the plasma concentration-time curve
Maximum plasma concentration (Cmax) | At the end of Cycle 1 (each cycle is 28 or 21 days)
  Maximum plasma concentration
Time to maximum plasma concentration (Tmax) | At the end of Cycle 1 (each cycle is 28 or 21 days)
  Time to maximum plasma concentration
Plasma half-life (t½) | At the end of Cycle 1 (each cycle is 28 or 21 days)
  Plasma half-life
Volume of distribution (Vd) | At the end of Cycle 1 (each cycle is 28 or 21 days)
  Volume of distribution
Plasma clearance (CL) | At the end of Cycle 1 (each cycle is 28 or 21 days)
  Plasma clearance
Cumulative urinary excretion rate of docetaxel prototypes | At the end of Cycle 1 (each cycle is 28 or 21 days)
  Cumulative urinary excretion rate of docetaxel prototypes
Preliminary identification of major metabolites in plasma and urine samples | At the end of Cycle 1 (each cycle is 28 or 21 days)
  Preliminary identification of major metabolites in plasma and urine samples

CONTACTS AND LOCATIONS:
Locations (1):
- Liu yunjiang, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No